CLINICAL TRIAL: NCT00840671
Title: A Prospective, Randomised, Placebo Controlled, Double Blind Trial About Safety and Efficacy of Combined Treatment With Alteplase (Rt-PA) and Cerebrolysin® in Acute Ischemic Hemispheric Stroke
Brief Title: Combined Treatment With Alteplase (Rt-PA) and Cerebrolysin® in Acute Ischemic Hemispheric Stroke
Acronym: CERE-LYSE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ever Neuro Pharma GmbH (Industry)
Collaborators: JSW-Research Forschungslabor GmbH, Parkring 12, 8074 Grambach (Unknown)
Responsible Party: Dr. Philipp Novak, EBEWE Neuro Pharma GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR040301; EudraCT-number: 2004-001729-11
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Stroke
Keywords: Cerebrolysin; Alteplase; Ischemic Stroke; Modified Rankin Scale; NIH Stroke Scale; Barthel Index; Glasgow Outcome Score
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — cerebrolysin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cerebrolysin (Experimental): Cerebrolysin, 30 ml/day as intravenous infusion, first infusion after completion of thrombolytic therapy. Daily infusion for 10 consecutive days.
  Interventions: Drug: Cerebrolysin
- 0.9% Saline Solution (Placebo Comparator): 0.9% Saline Solution, 30 ml/day as intravenous infusion, first infusion after completion of thrombolytic therapy. Daily infusion for 10 consecutive days.
  Interventions: Drug: 0.9% Saline Solution

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin, 30 ml/day as intravenous infusion, first infusion after completion of thrombolytic therapy. Daily infusion for 10 consecutive days.
  Arms: Cerebrolysin
Drug: 0.9% Saline Solution — 0.9% Saline Solution, 30 ml/day as intravenous infusion, first infusion after completion of thrombolytic therapy. Daily infusion for 10 consecutive days.
  Other Names: NaCl
  Arms: 0.9% Saline Solution

SUMMARY:
It should be shown that Cerebrolysin in combination with Alteplase, the medication that should recover the blood flow through the brain, is an effective and save medication to treat ischeamic stroke.

DETAILED DESCRIPTION:
The current trial should evaluate a combined treatment using Cerebrolysin immediately after thrombolysis to guarantee that the neurotrophic components are able to reach the endangered brain areas efficiently. An early start of treatment should guarantee rescue of most of the neurons reducing the overall damage.The study follows the design of pure thrombolytic trials to investigate, if the early neuroprotective treatment with Cerebrolysin is able to improve the overall outcome of patients at the day 90 evaluation visit. Due to the initial findings special emphasis will be also put on analysing the speed of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Female or male inpatients.
* Age: 18-80 years.
* If female, patient must not be pregnant
* Clinical diagnosis of ischemic stroke causing a measurable neurological deficit defined as impairment of language, motor function, cognition and/or gaze,vision or neglect. Ischemic stroke is defined as an event characterized by the sudden onset of an acute focal neurologic deficit presumed to be due to cerebral ischemia after CT scan excludes haemorrhage.
* Onset of symptoms within 3 hours prior to initiation of rt-PA administration.
* Stroke symptoms are to be present for at least 30 minutes and have not significantly improved before treatment. Symptoms must be distinguishable from an episode of generalized ischemia (i.e. syncope), seizure or migraine disorder.
* Patient is willing to participate voluntarily and to sign a written patient informed consent. Informed consent will be obtained from each patient or the subject's legally authorized representative or relatives, or deferred where applicable, according to the regulatory and legal requirements of the participating country.
* Patients who are unable to sign but who are able to understand the meaning of participation in the study may give an oral witnessed informed consent. These patients have to make clear undoubtful that they are willing to participate voluntarily and must be able to understand an explanation of the contents of the information sheet. A written consent has to be obtained as soon as possible.
* Willingness and ability to comply with the protocol.

Exclusion Criteria:

* Evidence of intracranial haemorrhage (ICH) on the CT-scan
* Violation of inclusion criteria not approved by clinical study director or study safety officer
* Failure to perform or to evaluate screening or baseline examinations
* Hospitalisation (except for study purposes) or change of concomitant medication 4 weeks prior to screening or during screening period
* Participation in another therapeutic clinical trial 3 months before baseline
* Patients with any history of prior stroke and concomitant diabetes
* Prior stroke within the last 3 months
* Platelet count of below 100x103/mm3
* Blood glucose <50 or >400 mg/dl (<2.77 or >22.15 mmol/L)
* Known haemorrhagic diathesis
* Manifest or recent severe or dangerous bleeding
* Known bacterial endocarditis, pericarditis
* Acute pancreatitis
* Documented ulcerative gastrointestinal disease during the last 3 months, oesophageal varices, arterial-aneurysm, arterial/venous malformation
* Neoplasm with increased bleeding risk
* Severe liver disease, including hepatic failure, cirrhosis, portal hypertension, oesaphageal varices) and active hepatitis
* Major surgery or significant trauma in past 3 months
* Lab values seriously abnormal, and/or more than 2 lab values abnormal not approved by clinical study director or study safety officer
* Serious drug allergies
* Hypersensitivity to one of the components of the drug
* Severe renal impairment
* Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, or aggressive management (IV medication) necessary to reduce BP to these limits
* Recent (less than 10 days) traumatic external heart massage, obstetrical delivery, recent puncture of a non-compressible blood-vessel (e.g. subclavian or jugular vein puncture)
* Chronic intoxication or chronic substance use disorder with pharmaceuticals, drugs, alcohol or industrial poisons
* Symptoms of ischemic attack began more than 3 hours prior to start of thrombolytic therapy or if time of symptom onset is unknown
* Minor neurological deficit or symptoms rapidly improving before start of infusion
* Severe stroke as assessed clinically (e.g. NIHSS >25) and/or by appropriate imaging techniques
* Epilepsy or epileptic seizure at onset of stroke
* Symptoms suggestive of subarachnoid haemorrhage, even if the CT-scan is normal
* Known history of or suspected intracranial haemorrhage
* Suspected subarachnoid haemorrhage or condition after subarachnoid hemorrhage from aneurysm
* Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
* Haemorrhagic retinopathy, e.g. in diabetes (vision disturbances may indicate haemorrhagic retinopathy)
* Administration of heparin within the previous 48 hours and a thromboplastin time exceeding the upper limit of normal for laboratory
* Patients receiving oral anticoagulants, e.g. warfarin sodium
* Special attention should be given to possible additive effects when used in conjunction with anti-depressants or MAO-inhibitors
* Cerebrolysin should not be mixed with balanced amino acid solutions in an infusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale score at day 90 (or earlier in the event of patient withdrawal). | Day 90

SECONDARY OUTCOMES:
NIH Stroke Scale Score 90 days after start of treatment (or earlier in the event of patient withdrawal). Actual score or change from baseline score analysed. | 90 days after start of treatment
Glasgow Outcome Score 90 days after start of treatment (or earlier in the event of patient withdrawal). Actual score or change from baseline score analysed. | 90 days after start of treatment
Barthel Index Score 90 days after start of treatment (or earlier in the event of patient withdrawal). Actual score or change from baseline score analysed. | 90 days after start of treatment
Responders classified according to Barthel Index Score ≥95, Glasgow Outcome Score 0-1, NIHSS change from baseline score, 8 point improvement or total score 0-1 or NIHSS Distal Motor Function Score 0-1. Responder rates across each scale analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Windisch, PhD, Study Director — JSW Research Forschungslabor GmbH; Wilfried Lang, MD, Principal Investigator — Krankenhaus der Barmherzigen Brüder, 1020 Wien
Locations (15):
- Austria (5):
  - Außenstelle Landesklinikum Donauregion Gugging, Gugging
  - Universitätsklinik Innsbruck, Dept. of Neurology, Innsbruck
  - LKH Klagenfurt, Abteilung für Neurologie, Klagenfurt
  - AKH Linz, Abteilung Neurologie & Psychiatrie, Linz
  - Krankenhaus der Barmherzigen Brüder/Abteilung für Neurologie, Vienna
- Croatia (4):
  - Klinicka Bolnicki Centar, Klinika za Nevrologiju, Rijeka
  - Clinical Hospital Split, Dept. of Neurology, Split
  - Medical School of Zagreb, Zagreb
  - University Hospital Sorrores Misericoridae, Zagreb
- Czechia (4):
  - St. Ann's Hospital, Dept. of Neurology, Brno
  - Clinic of Neurology, Faculty Hospital Ostrava, Ostrava
  - Blessed Mary Anthony Hospital, Dept. of Neurology, Ostrava Vitkovice
  - University Hospital Plzen, Pilsen
- University Hospital, Comenius University, Dept. of Neurology, Bratislava, Slovakia
- Clinical Hospital Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Lang W, Stadler CH, Poljakovic Z, Fleet D; Lyse Study Group. A prospective, randomized, placebo-controlled, double-blind trial about safety and efficacy of combined treatment with alteplase (rt-PA) and Cerebrolysin in acute ischaemic hemispheric stroke. Int J Stroke. 2013 Feb;8(2):95-104. doi: 10.1111/j.1747-4949.2012.00901.x. Epub 2012 Sep 26. PMID 23009193